CLINICAL TRIAL: NCT04729686
Title: The Pericapsular Nerve Block in Total Hip Arthroplasty: A Randomized, Controlled Trial
Brief Title: The Pericapsular Nerve Block in Total Hip Arthroplasty
Acronym: PENG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Rubin Institute for Advanced Orthopedics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1665162
Record Dates: First submitted 2020-12-22; First posted 2021-01-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy
Keywords: Total Hip Arthroplasty; Total Hip Replacement; Hip Arthroplasty; Hip Replacement; Postoperative Pain
MeSH Terms: conditions — Osteoarthritis, Hip; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pericapsular Nerve Block Group (Active Comparator): Pericapsular Nerve Block targets the anterior hip capsule by blocking the articular branches of the femoral nerve and accessory obturator nerve.
  Interventions: Drug: Pericapsular Nerve Block
- Fascia Iliaca Nerve Block Group (Active Comparator): Fascia Iliaca Nerve Block targets the space between the iliacus muscle and the fascia that overlies it (fascia iliaca), within which the femoral nerve and lateral femoral cutaneous nerve (LFCN) course.
  Interventions: Drug: Fascia Iliaca Nerve Block

INTERVENTIONS:
Drug: Pericapsular Nerve Block — Per Standard Institutional Practice
  Arms: Pericapsular Nerve Block Group
Drug: Fascia Iliaca Nerve Block — Per Standard Institutional Practice
  Arms: Fascia Iliaca Nerve Block Group

SUMMARY:
In order to continue progressing towards outpatient total hip arthroplasty (THA), methods to adequately manage postoperative pain is of paramount importance. The purpose of this study is to quantify the effectiveness of the pericapsular nerve block in total hip arthroplasty in comparison to the fascia iliaca nerve block.

DETAILED DESCRIPTION:
This is a single center, randomized, controlled trial in adult subjects undergoing total hip arthroplasty that will receive one of two different nerve block regimens for pain management as part of standard of care.

Effective pain control after surgery for total hip replacement is a critical element in patient recovery. Particularly, in the first few days, as majority of patients may experience significant pain. Improved pain management after surgery contributes to better healing, faster patient mobility, shortened hospital stays, and reduced healthcare costs. While pain management is an important factor in total hip replacement, pain after surgery has yet to be improved. Inadequate pain control can lead to delayed movement, thereby increasing the risk for complications such as blood clots in the legs (deep venous thrombosis - blood clots in your veins) with some patients developing blood clots in their lungs (pulmonary embolus). In addition to pain medications after surgery, nerve blocks such as the femoral or fascia iliaca, have been used as supporting therapy for pain management after a total hip replacement. While these nerve blocks are used on a regular basis, they do have limitations which can produce inconsistent results for pain control and use of pain medications after surgery. With no clear superior nerve block for total hip replacement, a new nerve block, called the pericapsular nerve group (PENG) block has emerged. It has demonstrated the ability to prolong pain relief and decrease the use of pain medications after surgery. Therefore, a randomized study comparing the PENG block to other blocks established within the anesthesia community (e.g., fascia iliaca block) will allow for providers to understand the capabilities this block has in the setting of a total hip replacement.

In addition to your normal standard clinical care, there will scheduled pre-operative, operative, 2-week, and 4-6 week follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Planned primary total hip arthroplasty with anterior (Smith-Peterson) approach
* ASA score of 1 to 3
* Indicated for one of the two nerve block groups
* Must be opioid naïve at screening as defined by the FDA - According to the Food and Drug Administration, opioid-tolerant patients were those currently receiving or who had previously received 60 mg PO morphine per day, 25 mcg transdermal fentanyl per hour, 30 mg PO oxycodone per day, 8 mg PO hydromorphone per day, 25 mg PO oxymorphone per day, 60 mg PO hydrocodone per day, or an equivalent dose of another opioid for a duration of one week or longer (16)

Exclusion Criteria:

* Current or previous diagnosis of "chronic pain"
* Opioid tolerant at time of screening (for a week or longer, at least 60 mg of morphine daily, or at least 30 mg of oral oxycodone daily, or at least 8 mg of oral hydromorphone daily or an equianalgesic dose of another opioid.)
* Diagnosis of ankylosing spondylitis
* Allergy to any potential medications utilized in any of the two groups
* Conversion of patient to general anesthesia intraoperatively
* Treatment with another investigational drug or other intervention for pain
* Any condition(s) or diagnosis, both physical or psychological, or physical exam finding in the opinion of the investigator that would precludes participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale (VAS) Score | Every 4 hours from end of surgery to 48 hours post surgery or discharge
  Score recorded by drawing a vertical line on a 100 mm horizontal line between "No Pain" (0 mm) and "Worst Pain" (100 mm)
Postoperative Opioid Consumption in mg | Surgery to 1 month post surgery
  Total opioid consumption will be recorded during postoperative period and at 1 month follow-up visit

SECONDARY OUTCOMES:
Time to first opioid medication | End of surgery 48 hours post-operation or discharge
Time to first ambulation | End of surgery to 48 hours post-operation or discharge
Distance upon first ambulation | 48 hours postoperative or discharge
Incidence of weakness and falls | End of surgery to 48 hours post-operation or discharge
Harris Hip Score | Last preoperative visit to four weeks post-operation
  10 question items measuring pain severity, function, absence of deformity, and range of motion. Scores range from 0-100 with higher scores representing better outcomes.
12 Item Short Form Health Survey Version 2 | Last preoperative visit to four weeks post-operation
  12 question items measuring health and well being as reported by the patient. 2 scores are calculated: 1) Physical Component Summary Score (PCS) and (2) Mental Health Component Summary Score (MCS) in which scores range from 0-100 with a score of zero indicating lowest level of health and 100 indicating the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Delanois, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States